CLINICAL TRIAL: NCT03754296
Title: Treatment of Acute Ischemic Stroke With CATCHVIEW Stent Retriever in Comparison to SOLITAIRE 2/FR - the TRUST Study - a Non-interventional, International, Multicenter, Prospective, Single-arm Study Based on an Objective Performance Criterion
Brief Title: Treatment of Acute Ischemic Stroke With CATCHVIEW Stent Retriever in Comparison to SOLITAIRE 2/FR
Acronym: TRUST
Status: Withdrawn | Type: Observational
Why Stopped: Strategic decision
Sponsor: Balt Extrusion (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-201703-CATCH
Record Dates: First submitted 2018-11-23; First posted 2018-11-27 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CATCHVIEW stent retriever
  Interventions: Device: CATCHVIEW

INTERVENTIONS:
Device: CATCHVIEW — Revascularization device

SUMMARY:
The TRUST study is a non-interventional, prospective, multicenter, international, single arm and non-inferiority study. It is designed to evaluate the efficacy and safety of mechanical thrombectomy of the CATCHVIEW device compared to SOLITAIRE 2/FR based on an objective performance criterion (OPC) defined with available and published clinical evidence gathered through the Solitaire clinical trials in the arterial revascularization of patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years old
* Clinical signs consistent with acute ischemic stroke
* Pre-stroke modified Rankin Score ≤ 1
* Patient able to be treated within 8 hours of onset of stroke symptoms and within 2 hours between qualifying imaging from CTA or MRA to groin puncture
* Initial NIHSS ≥ 6 and < 30 at the time of inclusion
* Arterial occlusion in the intracranial internal carotid, M1/M2 segment of the MCA, carotid terminus or tandem proximal ICA/MCA-M1 confirmed by CT or MR angiography that is accessible to the device
* Acute ischemic stroke where patient is ineligible for IV thrombolytic treatment or the treatment is contraindicated (e.g., patient presents beyond recommended time from symptom onset), or where patient has received IV thrombolytic therapy without partial or complete recanalization
* Primary use of the CATCHVIEW stent retriever for the procedure (decision of use is done independently and prior to the participation of the patient in the study)
* Life expectancy of at least 90 days
* Ability of the patient or legally authorized representative to provide a signed and dated informed consent form before the procedure. Where applicable, in case of medical emergency not allowing the patient to provide consent and unavailability of the legally authorized representative, a physician who does not take part in the study will sign the informed consent before the procedure. In any case, the patient or the legally authorized representative consent shall be requested as soon as possible after the procedure up until the discharge visit.

Exclusion Criteria:

Clinical exclusion criteria

* Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT or MRI scan is normal
* Suspicion of aortic dissection
* Patient with a co-morbid disease or condition that would confound the neurological and functional evaluations or compromise survival or ability to complete follow-up assessments within 90 days
* Known history of other arterial disease that would prevent the device from reaching the target vessel and/or preclude safe recovery of the device
* Patient who requires hemodialysis or peritoneal dialysis, or who have contraindication to an angiogram for whatever reason
* Serious sensitivity to radiographic contrast agents
* Sensitivity to nickel-titanium
* Patient with stenosis proximal to the thrombus site that may preclude safe recovery of the device
* Inability to reach the occlusion site
* Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR>3.0
* Current participation in an interventional investigation drug or device treatment study
* Pregnant women

Imaging exclusion criteria

* Baseline non-contrast CT or DWI MRI evidence of a moderate/large core deﬁned as extensive early ischemic changes of Alberta Stroke Program Early CT score (ASPECTS) < 6
* Imaging evidence that suggests, in the opinion of the Investigator, the patient is not appropriate for mechanical thrombectomy intervention (e.g. inability to navigate to target lesion, moderate/large infarct with poor collateral circulation, etc.)
* CT or MRI evidence of hemorrhage on presentation
* CT or MRI evidence of mass effect or intra-cranial tumour (except small meningioma)
* Imaging evidence of cerebral vasculitis
* CT or MRI showing an infarction core involving greater than 1/3 of the MCA territory (or in other territories > 100 cc of tissue) on presentation
* CT or MRI evidence of a basilar artery (BA) occlusion or posterior cerebral artery (PCA) occlusion

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with acute onset of stroke symptoms leading to significant clinical deficit in the setting of an angiographically proven occlusion of a proximal intracranial artery (intracranial internal carotid, middle cerebral M1 and/or M2 segments, carotid terminus or tandem proximal ICA/MCA-M1) who could have endovascular therapy (defined as the first pass with assigned study device) started within 8h of onset of stroke symptoms will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Score (mRS) | 90 days
  Proportion of patients achieving functional independence (mRS ≤ 2)

IPD SHARING:
Plan to Share IPD: No